CLINICAL TRIAL: NCT06490068
Title: An Open, Single-arm, Phase II Clinical Study to Evaluate the Efficacy and Safety of LTC004 in Combination With Toripalimab in Patients With Advanced Solid Tumors Resistant to First-line Immunotherapy
Brief Title: Study of LTC004 Combine With Toripalimab in Patient With Solid Tumors Resistant to Immunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTC004-204
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LTC004+Toripalimab (Experimental): Eligible subjects will receive LTC004 on day 1 of Week 1 and day 1 of week 3. Beginning at week 5, all subjects will receive LTC004 in combination with Toripalimab.
  Interventions: Drug: LTC004+Toripalimab

INTERVENTIONS:
Drug: LTC004+Toripalimab — LTC004 on D1 of Week 1 and D1 of week 3. IV,90μg/kg. Beginning at week 5, all subjects will receive LTC004 in combination with Toripalimab.
  LTC004:D3,iv,45μg/kg,Q3W. Toripalimab:D1,iv,240mg,Q3W.
  Other Names: LTC004 combine with Toripalimab

SUMMARY:
To evaluate the efficacy and safety of LTC004 in combination with Toripalimab in 10 patients with advanced solid tumors resistant to first-line immunotherapy, all eligible subjects will receive LTC004 on day 1 of Week 1 and day 1 of week 3. Beginning at week 5, all subjects will receive LTC004 in combination with Toripalimab regimen until disease progression, intolerance, informed withdrawal or up to 2 years of dosing, whichever occurred first.

DETAILED DESCRIPTION:
All eligible subjects will receive LTC004 on day 1 of Week 1 and day 1 of week 3. Beginning at week 5, all subjects will receive LTC004 in combination with Toripalimab regimen until disease progression, intolerance, informed withdrawal or up to 2 years of dosing, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years.
2. Locally advanced or metastatic solid tumors confirmed by pathology or cytology that cannot be surgically resected or can not be treated with radical concurrent chemoratherapy, and immune checkpoint inhibitor ± chemotherapy has become the standard first-line treatment, such as NSCLC, cervical cancer, head and neck squamous cell carcinoma, esophageal squamous cell carcinoma, etc. In addition, the patients had received no more than 1 line of systemic chemotherapy and no more than 1 line of systemic PD-1/PD-L1 inhibitor treatment at the same time or successively, and the treatment failed, and the previous PD-1/PD-L1 inhibitor treatment lasted more than 6 months, the best curative effect was CR/PR; No systemic antitumor therapy other than the above treatment was received (Note: if there is a second-line standard treatment, the second-line standard treatment is required to be completed before inclusion in this trial).
3. At least one measurable tumor lesion based on RECIST V1.1 criteria.
4. ECOG PS ≤1.
5. Expected survival ≥12 weeks.
6. Adequate organ function.
7. Patients, both females and males, of reproductive potential must agree to use adequate contraception during and for 6 months after the last infusion.
8. Understands and provides written informed consent and willing to follow the requirements specified in protocol.

Exclusion Criteria:

1. History of severe hypersensitivity reactions to other mAbs.
2. Untreated, unstable or uncontrolled central nervous system (CNS) metastases with following exceptions:A. Clinically stable MRI scans and no progressive or uncontrolled neurologic symptoms or signs for at least 4 weeks prior to the first study treatment.
3. Tumor invasion of vital arteries resulting in high risk of bleeding, significant risk of perforation or already formed fistulae.
4. Patients with uncontrolled pleural effusion, pericardial effusion or abdominal effusion as judged by the investigator at screening.
5. Patients with untreated or clinically symptomatic spinal cord compression that has not been controlled.
6. Previous antitumor regimens include immunotherapy such as LAG3, TIGIT, IL-2, IL-15, CD3-like immunoagonists, and other cellular therapies.
7. ≥2 malignant tumors within 5 years prior to first dose of drug.
8. irAE with ≥ grade 3 or discontinuation due to immunotherapy in the past.
9. Patients who have received any chemotherapy or anti-tumor monoclonal antibody drugs within 4 weeks prior to the first dose of study drug.small molecule targeted drugs within 2 weeks prior to the first dose of study drug; Chinese medicine therapy with clear anti-tumor indications in the package insert within 4 weeks prior to the first dose of study drug.
10. Severe infection, including but not limited to bacteremia requiring hospitalization and severe pneumonia, occurs within 4 weeks prior to the first medication; Active infection of grade CTCAE≥2 requiring treatment with systemic antibiotics was present within 2 weeks prior to the first dose.
11. The subject has active interstitial lung disease (ILD) or pneumonia; A history of needing hormones or other immunosuppressants to treat ILD or (non-infectious) pneumonia.
12. History of serious cardiovascular disease.
13. Active bleeding disorders, including gastrointestinal bleeding, as evidenced by vomiting of blood, profuse hemoptysis, or black stools, have occurred in the 6 months prior to enrollment.
14. Active hepatitis B,hepatitis C infection,syphilis infection, active tuberculosis.
15. Patients with active, or previous autoimmune disease with potential for recurrence.
16. Immunodeficiency diseases or history of such diseases, including a positive serologic test for human immunodeficiency virus (HIV).
17. Arterial/venous thrombotic events within 6 months prior to the first dose of the drug.
18. Those who received radical radiation therapy within 4 weeks prior to the first dose and those who received palliative radiation within 14 days prior to the first dose.
19. Use of live or attenuated vaccines within 4 weeks prior to the first dose,or anticipated need for live or attenuated vaccines during the study period.
20. Major surgery within 4 weeks prior to the first dose, anticipation of major surgery (other than surgery for diagnostic purposes) during the study period, or diagnostic or low-invasive surgery within 7 days prior to the first dose (excluded for puncture biopsies).
21. Adverse effects of prior antitumor therapy have not recovered to CTCAE version 5.0 grade rating ≤1.
22. Patients who have received a previous allogeneic bone marrow/hematopoietic stem cell transplant or solid organ transplant.
23. Pregnant and lactating women.
24. Subjects who in the judgment of the investigator, have a history of other serious systemic disease or are unfit to participate in this trial for any other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 12 months
  Antitumor efficacy of LTC004+Toripalimab treated patient with advanced solid tumors resistant to first-line immunotherapy

SECONDARY OUTCOMES:
DCR | up to 12 months
  Disease control rate of LTC004+Toripalimab treated patient with advanced solid tumors resistant to first-line immunotherapy
DOR | up to 12 months
  Duration of Response of LTC004+Toripalimab treated patient with advanced solid tumors resistant to first-line immunotherapy
PFS | up to 12 months
  Progression-Free Survival of LTC004+Toripalimab treated patient with advanced solid tumors resistant to first-line immunotherapy
OS | up to 12 months
  Overall Survival of LTC004+Toripalimab treated patient with advanced solid tumors resistant to first-line immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No